CLINICAL TRIAL: NCT06276530
Title: Impact of Surgical Approach on Adaptation of Posture-respiratory Coupling
Acronym: VaPosVent
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: APHP231036
Record Dates: First submitted 2023-12-19; First posted 2024-02-26 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Resectable Lung Non-Small Cell Carcinoma
Keywords: Posture-respiratory coupling,; Robotic-assisted thoracic surgery; Conventional thoracotomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Thoracotomy (Active Comparator): The patients in this group will have a major lung resection through a conventional postero-lateral thoracotomy.
  Interventions: Other: EOS imaging for musculoskeletal disorder; Other: Movement analysis by an optoelectronic camera.; Other: Stabilometric measurement by strength platform
- RATS (robotic-assisted thoracoscopic surgery) (Active Comparator): The patients in this group will have a major lung resection through a minimally invasive approach by RATS.
  Interventions: Other: EOS imaging for musculoskeletal disorder; Other: Movement analysis by an optoelectronic camera.; Other: Stabilometric measurement by strength platform

INTERVENTIONS:
Other: EOS imaging for musculoskeletal disorder — The patients will have a low radiation 2D/3D biplane imaging of the rib cage, and spine before and after surgery.
Other: Movement analysis by an optoelectronic camera. — Movement analysis by an optoelectronic camera before and after surgery.
Other: Stabilometric measurement by strength platform — Stabilometric measurement by strength platform before and after surgery.

SUMMARY:
This study aims to identify physiopathologic mechanisms related to surgical approaches during lobectomies for non-small cell lung cancer which can explain the better quality of life and the decrease of of post-operative complications in minimally invasive techniques (video-assisted thoracic surgery and robotic-assisted thoracic surgery) compared to conventional thoracotomy.

DETAILED DESCRIPTION:
In 2018, 46363 new cases of lung cancers have been diagnosed in France. It is the second most frequent cancer in men and the third most frequent cancer in women. It is the deadliest cancer in men and second deadliest cancer in women with 33117 deaths in 2018. The gold standard treatment is lobectomy with lymph node dissection in patients with a resectable tumor. The main surgical approach has long been conventional thoracotomy. It is associated with prolonged post-operative pain and discomfort because of rib spreading which injures the intercostal nerve and a costo-transverse disjunction. Moreover, in patients with narrowed intercostal space or restrictive syndrome, cher is a high risk of rib fracture associated. Alternative surgical approaches have been developed to reduce the pain and discomfort during a lobectomy. Minimally invasive approaches are mainly represented by video-assisted thoracic surgery (VATS) and robotic-assisted thoracic surgery (RATS). These approaches are characterized by the use of an endoscope during the whole procedure associated with specific instruments and the absence of rib spreading. With these technique, a similar disease-specific long-term survival is obtained compared to conventional thoracotomy. These techniques also reduce post-operative complications, post-operative acute and chronic pain and improve the quality of life. The discomfort and the decrease in quality of life comes from the pain related to the incision but could also come from the postural dysfunction , more frequent and severe after conventional thoracotomy. The physiopathology behind this postural dysfunction are not well known but seem to be related to partially to the mechanical alteration of the rib cage and partially and because of a mechanical dysfunction related to the diaphragm following the surgery. The rib cage is an important element of postural stability. The diaphragm has a key role in both breathing and posture. Alterations of these structures dedicated to stability and ventilation are potentially associated with central mechanisms which end up in an adaptation of posture-respiratory coupling. By comparing conventional thoracotomy and VATS, it has been shown that lobectomy by VATS is associated with less disruption in posture and posture-respiratory coupling compared to thoracotomy. But no data hast yet compared RATS and conventional thoracotomy. The investigators hypothesized that RATS would cause less disruption in the postural alignment, in the perception of verticality and posture-respiratory coupling index (in static position and by walking) compared to conventional thoracotomy. In this context, the investigators aim to compare the effects of conventional thoracotomy with RATS on the rib cage and the posture-respiratory coupling.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted for major lung resection
* Surgical approach by conventional postern-lateral thoracotomy
* Surgical approach by minimally invasive RATS

Exclusion Criteria:

- Extended lung resection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-03-25 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Thoracic kyphosis (T1- T12 angle) and vertical alignment head-pelvis and head- C7 vertebra (angle OD-HA and OD-C7) (EOS) | Assessment one week before surgery and 4 weeks surgery.
  Variation between pre- and post-operative measurement

SECONDARY OUTCOMES:
Width of rib cage (EOS) | Assessment one week before surgery and 4 weeks after surgery.
  Variation between pre- and post-operative measurement in centimeters
Rib cage volume (EOS) | Assessment one week before surgery and 4 weeks after surgery.
  Variation between pre- and post-operative measurement in Liter
" Umbrella "angle (EOS) | Assessment one week before surgery and 4 weeks after surgery
  Variation between pre- and post-operative measurement
Center of Pressure displacement (Optoelectronic system) | Assessment one week before surgery and 4 weeks after surgery
  Variation between pre- and post-operative measurement

CONTACTS AND LOCATIONS:
Overall Officials: Harry ETIENNE, M.D., PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Department of Thoracic and Vascular Surgery Tenon University Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Pujol JL, Thomas PA, Giraud P, Denis MG, Tretarre B, Roch B, Bommart S. Lung Cancer in France. J Thorac Oncol. 2021 Jan;16(1):21-29. doi: 10.1016/j.jtho.2020.09.012. No abstract available. PMID 33384058
- [Background] Postmus PE, Kerr KM, Oudkerk M, Senan S, Waller DA, Vansteenkiste J, Escriu C, Peters S; ESMO Guidelines Committee. Early and locally advanced non-small-cell lung cancer (NSCLC): ESMO Clinical Practice Guidelines for diagnosis, treatment and follow-up. Ann Oncol. 2017 Jul 1;28(suppl_4):iv1-iv21. doi: 10.1093/annonc/mdx222. No abstract available. PMID 28881918
- [Background] Cerfolio RJ, Price TN, Bryant AS, Sale Bass C, Bartolucci AA. Intracostal sutures decrease the pain of thoracotomy. Ann Thorac Surg. 2003 Aug;76(2):407-11; discussion 411-2. doi: 10.1016/s0003-4975(03)00447-8. PMID 12902074